CLINICAL TRIAL: NCT02185170
Title: Assessment of New Fluorescence Imagery Techniques Using Prostate Chips From Transurethral Resections.
Brief Title: DEPORRA-CoProst: Assessment of New Fluorescence Imagery Techniques Using Prostate Chips From Transurethral Resections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results of 5 first patients show that chips' cauterization interferes the signal
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire TIMC-IMAG (Other); FEMTO-ST Institute (Unknown); LLTech laboratory (Unknown); Clinical Investigation Center, Technological Innovation (Grenoble and Besancon) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 12 03
Record Dates: First submitted 2014-06-23; First posted 2014-07-09 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Medical Device; Fluorescence
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluorescence assesment (Experimental): All patients undergo a transurethral resection.
  There are four different steps in the study:
  * the first step: fresh prostatic tissue of 30 subjects will be use to asses the fluorescence signal and the entire chain,
  * the second step: fresh prostatic tissue of 10 subjects will be used to asses the immunolabelling protocol,
  * the third step: fresh prostatic tissue of 20 subjects will be used to asses the use of the FEMTO-ST institute medical device,
  * the four step: the fresh prostatic tissue from the 10 subjects of the second step will be evaluated to verify the preservation of morphological structure with the use of the Light-CT scanner.
  Interventions: Procedure: Trans-urethral resection; Device: Use of the FEMTO-ST institute medical device; Device: Use of the Light-CT scanner

INTERVENTIONS:
Procedure: Trans-urethral resection — All subjects of the study are going to have a trans-urethral resection of prostate.
Device: Use of the FEMTO-ST institute medical device — The FEMTO-ST institute medical device is use to detect prostatic and malignant tissue.
Device: Use of the Light-CT scanner — The Light-CT Scanner is use in the tissue structural observation

SUMMARY:
The aim of this study is divided in 4 different steps:

* the first step has two different purpose: assess the impact of the storage medium of fresh prostatic chips on fluorescence signal and adjust the entire chain (immunolabelling,counter-stain and imaging),
* the second step is the adaptation of immunolabelling protocol on histopathology slides, using fresh prostatic tissue,
* the third step is to validate the use of:

  1. the medical device created by the FEMTO-ST institute use for the detection of fluorescence signal on fresh tissue,
  2. the Light-CT scanner use for tissue structural observation.
* the four step is to check the preservation of morphological structure of tissue under the effect of laser excitation from the medical device.

ELIGIBILITY:
Inclusion Criteria:

* Male patient over 18 years old.
* Patient scheduled for trans-urethral resection of prostate with:

  1. prostate specific antigen (PSA) blood level ≤ 4 ng/ml and age > 80 years old
  2. a suspected prostate cancer after a digital rectal examination (DRE) and a PSA blood level > 50 ng/ml or an existing prostate cancer
* Patient affiliated to social security or beneficiary of such a regime.

Exclusion Criteria:

* Protected patient referred to in Articles L1121-6 to L1121-8 of the Code of Public Health

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Complete fluorescence measurement over each field of vision. | 1 day
  Determinate for the anti-PSMA antibody with Alexa Fluor 488 tracer, the ideal couple of antibody concentration/incubation time giving the highest immunofluorescent signal in the adjustment of fixed tissue sample protocol to fresh tissue sample protocol.

SECONDARY OUTCOMES:
Complete fluorescence measurement over each field of vision. | 1 day
  Determinate for the anti-PSMA antibody with R-Phycoerythrin tracer, the ideal couple of antibody concentration/incubation time giving the highest immunofluorescent signal in the adjustment of fixed tissue sample protocol to fresh tissue sample protocol.
Quality criteria of the structure of tissue (ordinal qualitative variables). | 1 day
  Verification of the preservation of morphological structure of tissue under the effect of laser excitation from the medical device.
Fluorescence measurements mean. | 1 day
  Validate the medical device from "FEMTO-ST institute" for the detection of fluorescence signals on fresh prostatic tissue.
Comparison of prostatic chips tissue architecture between the images from the Light-CT scanner and standard histopathology slides | 1 day
  Validate the Light-CT scanner from LLTech laboratory in the fresh prostatic tissue structural observation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Descotes, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Urology and Anatomopathology Department, Grenoble, France

REFERENCES:
- See also: Website of the Grenoble Clinical Investigation Center - Technological Innovation — http://www.cic-it-grenoble.fr
- See also: Website of the Techniques for biomedical engineering and complexity management - informatics, mathematics and applications - Grenoble laboratory — http://www-timc.imag.fr/
- See also: Website of FEMTO-ST — http://www.femto-st.fr/